CLINICAL TRIAL: NCT04650893
Title: The Effect of Intravenous Non-steroidal Anti-inflammatory Drugs and Intravenous Corticosteroids on the Likelihood of Dysphagia and Dysphonia Following Anterior Cervical Discectomy and Fusion
Brief Title: The Effect of IV NSAID's and Corticosteroids on Dysphasia and Dysphonia Following ASDF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor compliance with data collection - too many intervals.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0737-19-FB
Record Dates: First submitted 2020-11-12; First posted 2020-12-03 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Dysphagia; Dysphonia
MeSH Terms: conditions — Deglutition Disorders; Dysphonia

STUDY DESIGN:
Intervention Model Description: 25 patients into 3 separate arms.
Who Masked: Participant
Masking Description: Only patients will be masked from which cohort they were randomized into.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Control (Placebo Comparator): no steroid or non steroidal anti-inflammatory
  Interventions: Drug: Placebo
- Ketorolac (Active Comparator): one time dose of 30mg of IV Ketorolac at time of closure
  Interventions: Drug: Intravenous Ketorolac
- dexamethasone (Active Comparator): one time dose of 10mg of IV dexamethasone at the time of closure
  Interventions: Drug: Intravenous Dexamethasone

INTERVENTIONS:
Drug: Intravenous Ketorolac — To assess the efficacy of the meds for dysphagia and dysphonia following ACDF
  Arms: Ketorolac
Drug: Intravenous Dexamethasone — To assess the efficacy of the meds for dysphagia and dysphonia following ACDF
  Arms: dexamethasone
Drug: Placebo — Control
  Arms: Control

SUMMARY:
This study is to assess the efficacy of intra-operative intravenous non-steroidal anti-inflammatory drug (Ketorolac) versus intravenous (dexamethasone) administration on dysphagia and dysphonia after anterior cervical discectomy and fusion (ACDF).

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of two intra-operative, intravenous medications on dysphagia and dysphonia following anterior cervical discectomy and fusion (ACDF). The medications include Ketorolac, an anti-inflammatory versus dexamethasone, a corticosteroid. Eligibility criteria includes adults aged 19 years of age or older who are scheduled to undergo a ACDF for radiculopathy or myelopathy. Participants will be recruited for a prospective, randomized, single-blinded clinical drug study and randomized into three cohorts: (1) control (no steroid or non-steroidal anti-inflammatory (NSAID), (2) IV NSAID(1-time dose of 30mg of IV Ketorolac at time of closure), and (3) IV steroid (1-time dose of 10mg of IV dexamethasone at the time of closure. The primary outcome measures are patient questionnaires which include the EAT-10 and Bazaz classification for dysphagia and VHI-10 for dysphonia. In addition, the Neck Disability Index (NDI) and Visual Analogue Pain Scale (VAS) will also be collected. Research follow-up will be subject completed questionnaires to be collected pre-operatively and then post operation at day 1, 3 weeks, 6 weeks, 3 months, 6 months, and 1 year. Post operative questionnaires may be collected at time of patient follow-up in clinic, by phone or mail.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age and older
* Undergoing anterior cervical discectomy and fusion (ACDF) for radiculopathy or myelopathy
* No known allergies or sensitivities to steroid or non-steroidal medications

Exclusion Criteria:

* Procedure is being done for revision, trauma, infection or tumor
* Patients with known diagnosed metabolic diseases (diabetes, pancreatitis, gout, electrolyte imbalances, hypertension, hematological abnormalities including gastrointestinal bleeding...)
* Patients with known kidney disease or a creatinine level above the upper limit of normal >1.27

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Garvin, MD, Study Chair — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Lauritzen Outpatient Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated early, lack of compliance for follow-up intervals.
Groups:
- Ketorolac: one time dose of 30mg of IV Ketorolac at time of closure
  Intravenous Ketorolac: To assess the efficacy of the meds for dysphagia and dysphonia following anterior cervical discectomy and fusion (ACDF).
Period: Overall Study
Arm/Group | Control | Ketorolac | Dexamethasone
Started | 11 | 10 | 12
Completed | 0 | 0 | 1
Not Completed | 11 | 10 | 11
Not completed — Lost to Follow-up | 11 | 10 | 11

BASELINE CHARACTERISTICS:
Population: Baseline was less than desired due to closure of study because follow-up was poor.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Ketorolac | Dexamethasone | Total
Number analyzed (Participants) | 11 | 10 | 12 | 33
Age, Continuous [Mean (Full Range); unit: years] — Collection was questionnaires, no analysis completed due to poor patient compliance regarding follow-up. Population: Age data was not collected
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 5 | 16
  Male | 4 | 6 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 11 | 10 | 11 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Number of participants per study arm [Count of Participants; unit: Participants] | 11 | 10 | 12 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Moderate/Severe Bazaz Classification
Description: The Bazaz grading system (0-none; 1-Mild; 2-Moderate; 3-Severe) is used for dysphagia evaluation
Time Frame: one year
Measure: Number; unit: percentage of participants
Arm/Group | Control | Ketorolac | Dexamethasone
Number analyzed (Participants) | 5 | 5 | 4
percentage of participants | 20 | 20 | 0

2. Primary Outcome: Percentage of Patients With Severe Dysphagia Based on the Eating Assessment Tool (EAT-10)
Description: Percentage of patients with severe dysphagia based on the Eating Assessment Tool (EAT-10).Scores on the EAT-10 greater than 15 are indicative of severe dysphonia.
Time Frame: one year
Measure: Number; unit: percentage of participants
Arm/Group | Control | Ketorolac | Dexamethasone
Number analyzed (Participants) | 5 | 5 | 4
percentage of participants | 20 | 0 | 0

3. Secondary Outcome: Percentage of Patients With Clinically Significant Voice Handicap Index-10 (VHI-10).
Description: Scores on the VHI-10 greater than 11 are indicative of clinically significant dysphonia.
Time Frame: one year
Population: No placeholder numbers included; only one participant completed study.
Measure: Number; unit: percentage of participants
Arm/Group | Control | Ketorolac | Dexamethasone
Number analyzed (Participants) | 5 | 5 | 4
percentage of participants | 0 | 20 | 25

4. Secondary Outcome: Mean Neck Disability Index (NDI)
Description: The Neck Disability Index (NDI) is a 10 item pain intensity and daily activity questionnaire that measures daily limitations after cervical spine injury. There are 10 sections, and each section contains 6 statements.The statements are scored from 0 to 5, with 0 indicating no disability and 5 indicating complete disability.
  0: No disability or difficulty
  1. Mild disability or difficulty
  2. Moderate disability or difficulty
  3. Severe disability or difficulty
  4. Very severe disability or difficulty
  5. Complete disability or difficulty
  Total Score: The scores from each of the 10 sections are summed to calculate the total score. The maximum possible score is 50, which would indicate severe disability, while a score of 0 indicates no disability.
Time Frame: one year
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Control | Ketorolac | Dexamethasone
Number analyzed (Participants) | 5 | 5 | 4
score on a scale | 13.2 [1 to 28] | 16.2 [3 to 38] | 3.75 [0 to 9]

5. Other Pre Specified Outcome: Median Visual Analogue Scale for Neck Pain
Description: The Visual analogue scale is a line with numbers underneath it, with extremes marked "no pain" score of 0 (left) and the "worst pain imaginable" score of 10 (right).
Time Frame: one year
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Control | Ketorolac | Dexamethasone
Number analyzed (Participants) | 5 | 5 | 4
score on a scale | 2.6 [0 to 6] | 3.4 [0 to 6] | 1.75 [0 to 4]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Control | Ketorolac | Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT04650893/Prot_SAP_000.pdf